CLINICAL TRIAL: NCT05293327
Title: Immunohistochemical IMP3 and PCNA Expression as Diagnostic and Prognostic Markers in Laryngeal Squamous Cell Carcinoma in Sohag Governorate
Brief Title: IMP3 and PCNA Expression in Laryngeal Squamous Cell Carcinoma in Sohag Governorate
Acronym: IMP3PCNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Abdo Mohammed Abd El-latif, Assistant Lecturerof Pathology, Sohag University
Other Study IDs: Soh-Med-22-03-01
Record Dates: First submitted 2022-03-13; First posted 2022-03-24 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Laryngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laryngeal cancer is responsible for 2-5% of all new cancer cases worldwide. Squamous cell carcinoma of the larynx (LSCC) is the most common malignant tumor of the larynx, accounting for 85-90% of all laryngeal malignancies.

Despite significant therapeutic developments in recent decades, increases in patients' 5-year survival rates are still minimal , which is likely due to late-stage diagnosis and other complex factors. Therefore, to improve the outcome, timely diagnosis, selection of the most appropriate therapy, and an adequate follow-up approach is needed.

The insulin-like growth factor II m-RNA-binding protein 3 (IMP3) is a new biomarker that may be implicated in the carcinogenesis of various malignancies, including head and neck squamous cell carcinoma. IMP3 normally expressed in embryonic tissue but decreases after birth and is no longer detectable in adult tissue With the exception of a few tissues. As a result, IMP3 is expressed only in tumors and not in neighboring normal tissues.

Proliferating Cell Nuclear Antigen (PCNA) is a nuclear protein that acts as a cell proliferation marker. In most forms of solid malignancies, such as colorectal cancer and breast cancer, PCNA is closely linked to prognosis and survival.

In this study, hoping to improve diagnosis of LSCC and assess prognosis better by using both IMP3 and PCNA biomarkers. As IMP3 may have a role in cell growth and proliferation and PCNA is a marker of cell proliferation; studying the association between both markers in laryngeal carcinoma is recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Laryngeal resection (total or partial laryngectomy) and biopsies.
2. Complete clinical data.

Exclusion Criteria:

1. Patients with recurrence of the primary tumor.
2. Patients with a history of preoperative chemotherapy and/or radiotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Blocks obtained from laryngeal squamous cell carcinoma tissue previously extracted from patients treated in Sohag University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and prognosis of Laryngeal Squamous Cell Carcinoma | One or two days after staining sections with the markers
  Immunohistochemical Expression of IMP3 and PCNA in Laryngeal Squamous Cell Carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa AM Abd El-latif, Principal Investigator — Faculty of Medicine,Sohag University
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided